CLINICAL TRIAL: NCT03353077
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters on Squamous Cell Carcinoma
Brief Title: Alpha Radiation Emitters Device for the Treatment of Squamous Cell Carcinoma (DaRT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-SCC-000
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Skin Squamous Cell Carcinoma
Keywords: Skin SCC; Skin Carcinoma, Squamous

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alpha DaRT (Experimental): Alpha DaRT Seeds, Diffusing alpha-emitters Radiation Therapy.
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT

SUMMARY:
A unique approach for Skin Squamous Cell Carcinoma (SCC) treatment employing intratumoral diffusing alpha radiation emitter device

DETAILED DESCRIPTION:
This will be a prospective study, assessing the safety and effectiveness of intratumoral alpha radiation mediated treatment with Alpha DaRT seeds for the treatment of Skin Squamous Cell Carcinoma (SCC) tumors.

Treatment will be delivered through radioactive sources (Alpha DaRT seeds) inserted into the tumors in the skin. This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Lesions with histopathological diagnosis of squamous cell carcinoma will be studied.

Reduction in tumor size 30-45 days after DaRT insertion will be assessed. Safety will be assessed by the incidence, severity and frequency of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of skin squamous cell carcinoma before surgical removal of the tumor.
* Subjects with a tumor size ≤ 5 centimeters in the longest diameter (lesions without nodal spread).
* Subjects' age is over 18 years old.
* Subjects' ECOG Performance Status Scale is ≤ 2.
* Subjects' life expectancy is more than 6 months.
* Female subjects of childbearing age will have evidence of negative pregnancy test.
* Subjects are willing to sign an informed consent form.

Exclusion Criteria:

* Subject has a tumor with a maximal diameter > 5 centimeters.
* Subject has an ulcerative lesion.
* Subject has a tumor of Keratoacanthoma histology.
* Subjects' ECOG Performance Status Scale is ≥ 3.
* Patients with moribund diseases, e.g., autoimmune diseases, vasculitis, etc.
* Patients under immunosuppressive and/or corticosteroid treatment.
* Volunteers that participated in other studies in the past 30 days that might affect the evaluation of response or toxicity of DaRT.
* Pregnant women.
* Subjects not willing to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2019-07-14 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30-45 days post seed insertion
  The incidence, severity and frequency of all Adverse Events
Reduction in Tumor size | 30-45 days post seed insertion
  The reduction in tumor size 30-45 days after DaRT insertion

SECONDARY OUTCOMES:
Percent of NecroticTissue | 30-45 days post seed insertion
  Percent of necrotic tissue in the tumor 30-45 days after DaRT insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, Italy

IPD SHARING:
Plan to Share IPD: No